CLINICAL TRIAL: NCT02619227
Title: A Livelihood Intervention for Impoverished Women in Rural Uganda: Randomized Controlled Trial
Brief Title: A Livelihood Intervention for Impoverished Women in Rural Uganda
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mbarara University of Science and Technology (Other)
Responsible Party: Principal Investigator, Alexander Tsai, Assistant Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: MH096620-S3
Record Dates: First submitted 2015-08-15; First posted 2015-12-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Indigency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate treatment (Experimental): Participants will receive a livelihood intervention package consisting of a orientation and training and a loan package of chickens and associated implements to create poultry microenterprises
  Interventions: Other: Livelihood intervention
- Delayed treatment (No Intervention): Participants will receive no intervention but will be placed on a waitlist to receive the intervention after a 12-month delay.

INTERVENTIONS:
Other: Livelihood intervention — Participants will receive a livelihood intervention package consisting of a orientation and training and a loan package of chickens and associated implements to create poultry microenterprises.
  Arms: Immediate treatment

SUMMARY:
The objective of the study is to determine whether a livelihood intervention can improve economic and psychosocial wellbeing in rural Uganda.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-60 years (or emancipated minors aged 16-17 years) who live with at least one child under the age of 5 in the same household
* Women aged 18-60 years (or emancipated minors aged 16-17 years) who agree to participate in the livelihood intervention training program
* Women aged 18-60 years (or emancipated minors aged 16-17 years) who agree to participate in study data collection

Exclusion Criteria:

* Men
* Women who do not live in Nyakabare Parish
* Women under 18 years of age (if not emancipated minors) or older than 60 years of age
* Women who do not live with at least one child under the age of 5 in the same household
* Women who decline to participate in the livelihood intervention training program
* Women who decline to participate in study data collection
* Women who live in the same household as another study participant

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Household Food Insecurity Access Scale | 12 months
  Scale items range from 0 (never) to 3 (more than 10 days in the past month)
Hopkins Symptom Checklist Scale | 12 months
  Scale items range from 1 (not at all) to 4 (very much)

SECONDARY OUTCOMES:
Intimate Partner Violence Scale | 12 months
  Experience (yes/no) of 12 different forms of emotional, sexual, or physical victimization by an intimate partner (range 0-12)
Norms about Intimate Partner Violence Scale | 12 months
  Agreement (yes/no) with 5 different statements about the acceptability of intimate partner violence under 5 different scenarios (range, 0-5)
Self-Reported Health Scale | 12 months
  Scale item ranges from 1 (very bad) to 4 (very good)
Decision Making Power Scale | 12 months
  Primary decision making (yes/no) on household expenditures in 7 different categories: food, livestock, health care, transport, social, educational, other household (range, 0-7)
Social Integration Scale | 12 months
  Frequency of participation in 11 different community groups: vocational, positive living, local council, water, village health, agricultural extension, savings, religious, women's, gardening (range, 0-11)
Social Capital Scale | 12 months
  Agreement (yes/no) with 4 questions about social trust and social cohesion (range, 0-4)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander C Tsai, MD, PhD, Principal Investigator — Massachusetts General Hospital; Bernard Kakuhikire, MBA, Principal Investigator — Mbarara University of Science and Technology
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda

REFERENCES:
- [Derived] Weil AA, Debela MD, Muyanja DM, Kakuhikire B, Baguma C, Bangsberg DR, Tsai AC, Lai PS. Gut carriage of antimicrobial resistance genes in women exposed to small-scale poultry farms in rural Uganda: A feasibility study. PLoS One. 2020 Jun 11;15(6):e0229699. doi: 10.1371/journal.pone.0229699. eCollection 2020. PMID 32525954